CLINICAL TRIAL: NCT05185271
Title: Adopting Dyad-focused Strategy Training to Stroke Survivors and Their Caregivers: Intervention Development and a Feasibility Study
Brief Title: Adopting Dyad-focused Strategy Training to Stroke Survivors and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Feng-Hang Chang, Professor, Taipei Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N202106087
Record Dates: First submitted 2021-12-10; First posted 2022-01-11 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Stroke
Keywords: Caregiver; Stroke; Rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dyad- focused strategy training intervention (Experimental): The dyad-focused strategy training intervention protocol will be developed to help dyads manage the needs that they have as transitioning to the community.
  The following theoretical frameworks and guidelines will be used to guide the development of the intervention: (1) the strategy training guideline outlined by Skidmore et al; (2) Bodenmann's framework of dyadic coping; and (3) Self-efficacy theory.
  Interventions: Behavioral: Dyad-focused strategy training

INTERVENTIONS:
Behavioral: Dyad-focused strategy training — Rehabilitation therapists will be hired to deliver the intervention to the stroke survivors-caregiver dyads on a one-to-two base. The therapist will ask the dyad to identify their shared goals and provide them the global strategy "Goal-Plan-Do-Check" (also called guided discovery strategy), which involves (1) setting a goal to address the barriers, (2) developing a plan to address the goal, (3) doing the plan, and (4) checking if the plan worked or required revising. This procedure will be repeated iteratively until the dyad's goal is met, and the next goal can be moved on to.

SUMMARY:
The purpose of this study is to develop a dyad-focused intervention built upon the theoretical tenets of strategy training to help prepare stroke survivors and their caregivers to transit to community living. The study will involve two phases.

In phase one, the intervention protocol will be developed through literature review, expert panel meeting, and focus groups with rehabilitation therapists, stroke survivors, and caregivers. In phase two, a feasibility study will be conducted to evaluate the acceptability and suitability of this newly-developed intervention and outcome measures to stroke survivor-caregiver dyads.

A mixed-methods (quantitative and qualitative) design, including a repeated measures design, will be used in this feasibility study. Fifteen to twenty stroke survivor-caregiver dyads are expected to be recruited.

The participants will receive the dyad-focused strategy training intervention using the developed intervention protocol. Standardized assessments will be used to assess dyadic outcomes at baseline, post-intervention, and 3-month and 6-month follow-ups. Quantitative data will be analyzed descriptively.

DETAILED DESCRIPTION:
Stroke is the leading cause of death and adult disability. Transitioning from hospital to home is a challenging process for stroke survivors and their families, leading to frustration and adverse health outcomes for survivors and caregivers. To address both the survivor and caregiver needs, dyad-focused interventions are necessary to be implemented in the transitioning process. However, very few interventions were designed to address the needs of the dyad and place an equal emphasis on both survivors' and caregivers' outcomes.

The purpose of this study is to develop a dyad-focused intervention built upon the theoretical tenets of strategy training to help prepare stroke survivors and their caregivers to transit to community living. The study will involve two phases. In phase one, the intervention protocol will be developed through literature review, expert panel meeting, and focus groups with rehabilitation therapists, stroke survivors, and caregivers. In phase two, a feasibility study will be conducted to evaluate the acceptability and suitability of this newly-developed intervention and outcome measures to stroke survivor-caregiver dyads.

A mixed-methods (quantitative and qualitative) design, including a repeated measures design, will be used in this feasibility study. Fifteen to twenty stroke survivor-caregiver dyads are expected to be recruited. Adult stroke survivors who have been diagnosed with stroke, are about to be discharged from inpatient wards to home or has been discharged home within the past 3 months, have an identified adult caregiver who provides care or assistance of any kind and taking responsibility for the survivor and is available to participate in the intervention sessions with the survivor will be eligible to participate in the study. These participants will receive the dyad-focused strategy training intervention using the developed intervention protocol. Standardized assessments will be used to assess dyadic outcomes such as goal attainment, quality of life, self-efficacy, participation, depressive symptoms, and survivor-caregiver relationship at baseline, post-intervention, and 3-month and 6-month follow-ups. The feasibility indicators, such as recruitment rates and intervention attendance and adherence, will be evaluated by questionnaires, field notes, and qualitative interviews after the interventions are completed.

Quantitative data will be analyzed descriptively; while data obtained from the outcome measures will be examined using Wilcoxon signed rank test and effect size (r) to compare the differences between the pre- and post-intervention scores. Qualitative data will be analyzed using thematic analysis method.

ELIGIBILITY:
Inclusion Criteria:

Stroke survivors include that the survivor:

1. ages 20 years and older;
2. has been diagnosed with stroke;
3. speaks Mandarin;
4. is about to be discharged from inpatient wards to home or has been discharged home within the past 3 months;
5. has an identified primary caregiver;
6. is able to provide informed consent.

Caregivers include that the caregiver:

1. ages 20 years and older;
2. speaks Mandarin;
3. is the primary caregiver recognized by the survivor (living with the survivor or providing daily care to the survivor for at least 10 hours per week);
4. is available to participate in the intervention sessions with the survivor;
5. is able to provide informed consent.

Exclusion Criteria:

1. requires significant medical treatment (e.g., chemotherapy, radiation therapy, or hemo/peritoneal dialysis) that may impede them from participating in the study;
2. has severe aphasia;
3. is unable to participate in a 1-hour discussion session;
4. has a diagnosis of dementia, major depressive disorder, substance use or other psychiatric disorders that may impede them from continually participating in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Rehabilitation Participation Scale (PRPS) | During intervention, up to 2 months
  The PRPS, a clinician-rated instrument, measures patients' participation on a 6-point Likert-type scale. A higher point reflects better participation in each intervention session.
Client Satisfaction Questionnaire (CSQ) | Immediately after intervention
  The CSQ is an 8-item measure of client satisfaction with the intervention. It allows clients to rate on a 4-point scale where 1 represents "Not at all" and 4 represents "Extremely ." A higher score reflects higher satisfaction and acceptability of the intervention.
Qualitative data | After intervention
  Qualitative data will be collected through field notes taken by therapists after each intervention session and in-person qualitative interviews with participants and their therapists using semi-structured questionnaires.

SECONDARY OUTCOMES:
Goal Attainment Scaling (GAS) | Change from baseline to immediately post-intervention
  GAS is a method of scoring the extent to which patients' individual goals are achieved in intervention. If the patient achieves the expected level, this is scored at 0. If they achieve a better than expected outcome, this is scored at +1 (somewhat better) or +2 (much better). If they achieve a worse than expected outcome this is scored at -1 (partially achieved), -2 (No change) or -3 (much worse). Goals will be weighted to take account of the relative importance of the goal to the individual and/or the anticipated difficulty of achieving it.
World Health Organization Quality of Life (WHOQOL-Brief) Taiwan version | Change from baseline to immediately post-intervention
  The WHOQOL-BREF (Taiwan ver.) is a self-administered questionnaire comprising 28 questions on individuals' perceptions of their health and well-being over the previous two weeks. Responses to questions are on a 1-5 Likert scale where 1 represents "disagree" or "not at all" and 5 represents "completely agree" or "extremely".
World Health Organization Quality of Life (WHOQOL-Brief) Taiwan version | Change from post-intervention to 3-month follow-up
  The WHOQOL-BREF (Taiwan ver.) is a self-administered questionnaire comprising 28 questions on individuals' perceptions of their health and well-being over the previous two weeks. Responses to questions are on a 1-5 Likert scale where 1 represents "disagree" or "not at all" and 5 represents "completely agree" or "extremely".
World Health Organization Quality of Life (WHOQOL-Brief) Taiwan version | Change from 3-month to 6-month follow-up
  The WHOQOL-BREF (Taiwan ver.) is a self-administered questionnaire comprising 28 questions on individuals' perceptions of their health and well-being over the previous two weeks. Responses to questions are on a 1-5 Likert scale where 1 represents "disagree" or "not at all" and 5 represents "completely agree" or "extremely".
General Self-Efficacy Scale (GSES) | Change from baseline to immediately post-intervention
  The GSES, sometimes seen as GSE, is a 10-item psychometric scale created to assess perceived self-efficacy regarding coping and adaptation abilities in daily activities and isolated stressful events. Responses to questions are on a 1-4 Likert scale where 1 represents "Not at all true" and 4 represents "Exactly true."
General Self-Efficacy Scale (GSES) | Change from post-intervention to 3-month follow-up
  The GSES, sometimes seen as GSE, is a 10-item psychometric scale created to assess perceived self-efficacy regarding coping and adaptation abilities in daily activities and isolated stressful events. Responses to questions are on a 1-4 Likert scale where 1 represents "Not at all true" and 4 represents "Exactly true."
General Self-Efficacy Scale (GSES) | Change from 3-month to 6-month follow-up
  The GSES, sometimes seen as GSE, is a 10-item psychometric scale created to assess perceived self-efficacy regarding coping and adaptation abilities in daily activities and isolated stressful events. Responses to questions are on a 1-4 Likert scale where 1 represents "Not at all true" and 4 represents "Exactly true."
Participation Measure- 3 Domains, 4 Dimensions (PM-3D4D) | Change from baseline to immediately post-intervention
  The PM-3D4D is a 19-item measure that was designed to evaluate three domains of participation: Productivity, Social, and Community. Respondents are asked to rate each item on four dimensions: (1) 'Diversity of participation' (yes [1] vs. no [0]); (2) 'Frequency'(5- and 7-point scales, from "never" to "everyday or almost everyday"); (3) 'Desire for change' (yes [1] vs. no[0]); and (4) 'Perceived difficulty' (4-point scale, from "very difficult" [1] to "not difficult at all" [4]). Each dimensional score of the PM-3D4D can be separately summed for each domain. Psychometric properties of the PM-3D4D were established in rehabilitation populations.
Participation Measure- 3 Domains, 4 Dimensions (PM-3D4D) | Change from post-intervention to 3-month follow-up
  The PM-3D4D is a 19-item measure that was designed to evaluate three domains of participation: Productivity, Social, and Community. Respondents are asked to rate each item on four dimensions: (1) 'Diversity of participation' (yes [1] vs. no [0]); (2) 'Frequency'(5- and 7-point scales, from "never" to "everyday or almost everyday"); (3) 'Desire for change' (yes [1] vs. no[0]); and (4) 'Perceived difficulty' (4-point scale, from "very difficult" [1] to "not difficult at all" [4]). Each dimensional score of the PM-3D4D can be separately summed for each domain. Psychometric properties of the PM-3D4D were established in rehabilitation populations.
Participation Measure- 3 Domains, 4 Dimensions (PM-3D4D) | Change from 3-month to 6-month follow-up
  The PM-3D4D is a 19-item measure that was designed to evaluate three domains of participation: Productivity, Social, and Community. Respondents are asked to rate each item on four dimensions: (1) 'Diversity of participation' (yes [1] vs. no [0]); (2) 'Frequency'(5- and 7-point scales, from "never" to "everyday or almost everyday"); (3) 'Desire for change' (yes [1] vs. no[0]); and (4) 'Perceived difficulty' (4-point scale, from "very difficult" [1] to "not difficult at all" [4]). Each dimensional score of the PM-3D4D can be separately summed for each domain. Psychometric properties of the PM-3D4D were established in rehabilitation populations.
Hospital Anxiety and Depression Scale (HADS) | Change from baseline to immediately post-intervention
  The HADS is a fourteen-item scale that generates seven items related to anxiety and seven related to depression. Each item on the questionnaire is scored from 0-3, which means that a person can score between 0 and 21 for either anxiety or depression. Higher scores mean a worse outcome.
Hospital Anxiety and Depression Scale (HADS) | Change from post-intervention to 3-month follow-up
  The HADS is a fourteen-item scale that generates seven items related to anxiety and seven related to depression. Each item on the questionnaire is scored from 0-3, which means that a person can score between 0 and 21 for either anxiety or depression. Higher scores mean a worse outcome.
Hospital Anxiety and Depression Scale (HADS) | Change from 3-month to 6-month follow-up
  The HADS is a fourteen-item scale that generates seven items related to anxiety and seven related to depression. Each item on the questionnaire is scored from 0-3, which means that a person can score between 0 and 21 for either anxiety or depression. Higher scores mean a worse outcome.
Dyadic Relationship Scale (DRS) | Change from baseline to immediately post-intervention
  The DRS measures negative and positive dyadic interactions from the perspective of both patients and the family caregivers. The patient version (10 items) and the caregiver version (11 items) have two subscales: dyadic strain and positive dyadic interaction. Each item included a four-option response (1 = strongly disagree, 2 = disagree, 3 = agree, 4 = strongly agree). Higher scores on each of these scales indicate higher strain levels and positive interaction, respectively.
Dyadic Relationship Scale (DRS) | Change from post-intervention to 3-month follow-up
  The DRS measures negative and positive dyadic interactions from the perspective of both patients and the family caregivers. The patient version (10 items) and the caregiver version (11 items) have two subscales: dyadic strain and positive dyadic interaction. Each item included a four-option response (1 = strongly disagree, 2 = disagree, 3 = agree, 4 = strongly agree). Higher scores on each of these scales indicate higher strain levels and positive interaction, respectively.
Dyadic Relationship Scale (DRS) | Change from 3-month to 6-month follow-up
  The DRS measures negative and positive dyadic interactions from the perspective of both patients and the family caregivers. The patient version (10 items) and the caregiver version (11 items) have two subscales: dyadic strain and positive dyadic interaction. Each item included a four-option response (1 = strongly disagree, 2 = disagree, 3 = agree, 4 = strongly agree). Higher scores on each of these scales indicate higher strain levels and positive interaction, respectively.
Activity Measure for Post-Acute Care (AM-PAC) Short Forms | Change from baseline to immediately post-intervention
  The AM-PAC consists of three subscales that assess three activity domains: basic mobility, daily activity, and applied cognitive. The inpatient short consists of 6 items per domain, and the outpatient short consists of 15-19 per domain. Each item asks the respondent to rate the difficulty of performing specified activities using a 4-point scale. The summary scores for each subscale will be transformed into standardized scores on the t-score scale.
Activity Measure for Post-Acute Care (AM-PAC) Short Forms | Change from post-intervention to 3-month follow-up
  The AM-PAC consists of three subscales that assess three activity domains: basic mobility, daily activity, and applied cognitive. The inpatient short consists of 6 items per domain, and the outpatient short consists of 15-19 per domain. Each item asks the respondent to rate the difficulty of performing specified activities using a 4-point scale. The summary scores for each subscale will be transformed into standardized scores on the t-score scale.
Activity Measure for Post-Acute Care Short Forms | Change from 3-month to 6-month follow-up
  The AM-PAC consists of three subscales that assess three activity domains: basic mobility, daily activity, and applied cognitive. The inpatient short consists of 6 items per domain, and the outpatient short consists of 15-19 per domain. Each item asks the respondent to rate the difficulty of performing specified activities using a 4-point scale. The summary scores for each subscale will be transformed into standardized scores on the t-score scale.
Trail-Making Test (TMT A and B) | Change from baseline to immediately post-intervention
  The TMT test measures sustained attention, sequencing, mental flexibility, and visual tracking. TMT-A requires the individual to link in an ascending order a series of 25 numbered circles distributed randomly on a test paper as quickly as possible. TMT-B is similar, although it requires the individual to link switching alternatively between a set of numbers (1-13) and a set of letters (A-L) in ascending order (1-A-2-B-3-C...). The Time to complete TMT A and B will be calculated, in which a longer completion time will indicate a poorer outcome.
Trail-Making Test (TMT A and B) | Change from post-intervention to 3-month follow-up
  The TMT test measures sustained attention, sequencing, mental flexibility, and visual tracking. TMT-A requires the individual to link in an ascending order a series of 25 numbered circles distributed randomly on a test paper as quickly as possible. TMT-B is similar, although it requires the individual to link switching alternatively between a set of numbers (1-13) and a set of letters (A-L) in ascending order (1-A-2-B-3-C...). The Time to complete TMT A and B will be calculated, in which a longer completion time will indicate a poorer outcome.
Trail-Making Test (TMT A and B) | Change from 3-month to 6-month follow-up
  The TMT test measures sustained attention, sequencing, mental flexibility, and visual tracking. TMT-A requires the individual to link in an ascending order a series of 25 numbered circles distributed randomly on a test paper as quickly as possible. TMT-B is similar, although it requires the individual to link switching alternatively between a set of numbers (1-13) and a set of letters (A-L) in ascending order (1-A-2-B-3-C...). The Time to complete TMT A and B will be calculated, in which a longer completion time will indicate a poorer outcome.
Stroop Test | Change from baseline to immediately post-intervention
  The Stroop test assesses the ability to inhibit cognitive interference that occurs when processing a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute. Participants will be asked to read out the word's ink color as accurately as soon as possible. The ink color of the word could be congruent or incongruent with the written color name. Each participant's time to complete the task will be calculated and recorded.
Stroop Test | Change from post-intervention to 3-month follow-up
  The Stroop test assesses the ability to inhibit cognitive interference that occurs when processing a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute. Participants will be asked to read out the word's ink color as accurately as soon as possible. The ink color of the word could be congruent or incongruent with the written color name. Each participant's time to complete the task will be calculated and recorded.
Stroop Test | Change from 3-month to 6-month follow-up
  The Stroop test assesses the ability to inhibit cognitive interference that occurs when processing a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute. Participants will be asked to read out the word's ink color as accurately as soon as possible. The ink color of the word could be congruent or incongruent with the written color name. Each participant's time to complete the task will be calculated and recorded.
Montreal Cognitive Assessment (MoCA) | Change from baseline to immediately post-intervention
  MoCA is a 30-question test. It checks different cognitive or thinking abilities to help people quickly assess a patient's cognitive health.
  The score ranges from 0 to 30. A score of 26 and higher is considered normal.
Montreal Cognitive Assessment (MoCA) | Change from post-intervention to 3-month follow-up
  MoCA is a 30-question test. It checks different cognitive or thinking abilities to help people quickly assess a patient's cognitive health.
  The score ranges from 0 to 30. A score of 26 and higher is considered normal.
Montreal Cognitive Assessment (MoCA) | Change from 3-month to 6-month follow-up
  MoCA is a 30-question test. It checks different cognitive or thinking abilities to help people quickly assess a patient's cognitive health.
  The score ranges from 0 to 30. A score of 26 and higher is considered normal.
Preparedness for Caregiving Scale (CPS) | Change from baseline to immediately post-intervention
  The CPS is a caregiver self-rated instrument that consists of eight items that ask caregivers how well prepared they believe they are for multiple domains of caregiving. Responses rate on a 5 point scale with scores ranging from 0 (not at all prepared) to 4 (very well prepared). The scale is scored by calculating the mean of all items answered with a score range of 0 to 4. The higher the score, the more prepared the caregiver feels for caregiving; the lower the score, the less prepared the caregiver feels.
Preparedness for Caregiving Scale (CPS) | Change from post-intervention to 3-month follow-up
  The CPS is a caregiver self-rated instrument that consists of eight items that ask caregivers how well prepared they believe they are for multiple domains of caregiving. Responses rate on a 5 point scale with scores ranging from 0 (not at all prepared) to 4 (very well prepared). The scale is scored by calculating the mean of all items answered with a score range of 0 to 4. The higher the score, the more prepared the caregiver feels for caregiving; the lower the score, the less prepared the caregiver feels.
Preparedness for Caregiving Scale (CPS) | Change from 3-month to 6-month follow-up
  The CPS is a caregiver self-rated instrument that consists of eight items that ask caregivers how well prepared they believe they are for multiple domains of caregiving. Responses rate on a 5 point scale with scores ranging from 0 (not at all prepared) to 4 (very well prepared). The scale is scored by calculating the mean of all items answered with a score range of 0 to 4. The higher the score, the more prepared the caregiver feels for caregiving; the lower the score, the less prepared the caregiver feels.
The Zarit Burden Interview (ZBI) | Change from baseline to immediately post-intervention
  The ZBI, a caregiver self-report measure, contains 22 items to assess the caring burden. Each item on the interview is a statement which the caregiver is asked to endorse using a 5-point scale. Response options range from 0 (Never) to 4 (Nearly Always). A higher score means a worse outcome.
The Zarit Burden Interview (ZBI) | Change from post-intervention to 3-month follow-up
  The ZBI, a caregiver self-report measure, contains 22 items to assess the caring burden. Each item on the interview is a statement which the caregiver is asked to endorse using a 5-point scale. Response options range from 0 (Never) to 4 (Nearly Always). A higher score means a worse outcome.
The Zarit Burden Interview (ZBI) | Change from 3-month to 6-month follow-up
  The ZBI, a caregiver self-report measure, contains 22 items to assess the caring burden. Each item on the interview is a statement which the caregiver is asked to endorse using a 5-point scale. Response options range from 0 (Never) to 4 (Nearly Always). A higher score means a worse outcome.

OTHER OUTCOMES:
National Institutes of Health Stroke Scale | At baseline
  The NIHSS is a 15-item neurologic examination stroke scale used to evaluate the effect of stroke on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. The score will be calculated to quantify stroke severity.
Modified Rankin Scale (MRS) | Change from baseline to immediately post-intervention
  The MRS measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale runs from 0-6 ( Health without symptoms to death).
Modified Rankin Scale (MRS) | Change from post-intervention to 3-month follow-up
  The MRS measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale runs from 0-6 ( Health without symptoms to death).
Modified Rankin Scale (MRS) | Change from 3-month to 6-month follow-up
  The MRS measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale runs from 0-6 ( Health without symptoms to death).
HEAL Positive Outlook questionnaire (Short form) | Change from baseline to immediately post-intervention
  HEAL positive outlook questionnaire is a self-report measure that assesses participants' positive attitudes. The short form contains six items. Responses to questions are on a 1-5 Likert scale where 1 represents "Not at all" and 4 represents "Extremely ."
HEAL Positive Outlook questionnaire (Short form) | Change from post-intervention to 3-month follow-up
  HEAL positive outlook questionnaire is a self-report measure that assesses participants' positive attitudes. The short form contains six items. Responses to questions are on a 1-5 Likert scale where 1 represents "Not at all" and 4 represents "Extremely ."
HEAL Positive Outlook questionnaire (Short form) | Change from 3-month to 6-month follow-up
  HEAL positive outlook questionnaire is a self-report measure that assesses participants' positive attitudes. The short form contains six items. Responses to questions are on a 1-5 Likert scale where 1 represents "Not at all" and 4 represents "Extremely ."
HEAL Patient-Provider Connection | After the fifth intervention session, an average of 3 weeks
  HEAL Patient-Provider Connection is a self-report measure that assesses the relationship between a patient and a health care provider. It contains seven items. Responses to questions are on a 1-5 Likert scale where 1 represents "Not at all" and 4 represents "Extremely ."
HEAL Treatment Expectancy | After the first intervention session, an average of 1 week
  HEAL Treatment Expectancy is a self-report measure that assesses patients' expectations from the intervention. It contains six items. Responses to questions are on a 1-5 Likert scale where 1 represents "Not at all" and 4 represents "Extremely ."

CONTACTS AND LOCATIONS:
Overall Officials: Feng-Hang Chang, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Juengst SB, Osborne CL, Holavanahalli R, Silva V, Kew CL, Nabasny A, Bell KR. Feasibility Study of Problem-Solving Training for Care Partners of Adults With Traumatic Brain Injury, Spinal Cord Injury, Burn Injury, or Stroke During the Inpatient Hospital Stay. Arch Rehabil Res Clin Transl. 2019 Jun 27;1(3-4):100009. doi: 10.1016/j.arrct.2019.100009. eCollection 2019 Dec. PMID 33543049
- [Background] Haley WE, Roth DL, Hovater M, Clay OJ. Long-term impact of stroke on family caregiver well-being: a population-based case-control study. Neurology. 2015 Mar 31;84(13):1323-9. doi: 10.1212/WNL.0000000000001418. Epub 2015 Mar 4. PMID 25740862
- [Background] Moon M. The Unprepared Caregiver. Gerontologist. 2017 Feb;57(1):26-31. doi: 10.1093/geront/gnw080. Epub 2016 Apr 21. PMID 27106827
- [Background] Hare R, Rogers H, Lester H, McManus R, Mant J. What do stroke patients and their carers want from community services? Fam Pract. 2006 Feb;23(1):131-6. doi: 10.1093/fampra/cmi098. Epub 2005 Nov 24. PMID 16308328
- [Background] Duncan PW, Zorowitz R, Bates B, Choi JY, Glasberg JJ, Graham GD, Katz RC, Lamberty K, Reker D. Management of Adult Stroke Rehabilitation Care: a clinical practice guideline. Stroke. 2005 Sep;36(9):e100-43. doi: 10.1161/01.STR.0000180861.54180.FF. No abstract available. PMID 16120836
- [Background] Miller EL, Murray L, Richards L, Zorowitz RD, Bakas T, Clark P, Billinger SA; American Heart Association Council on Cardiovascular Nursing and the Stroke Council. Comprehensive overview of nursing and interdisciplinary rehabilitation care of the stroke patient: a scientific statement from the American Heart Association. Stroke. 2010 Oct;41(10):2402-48. doi: 10.1161/STR.0b013e3181e7512b. Epub 2010 Sep 2. No abstract available. PMID 20813995
- [Background] Jolly M, Thakkar A, Mikolaitis RA, Block JA. Caregiving, dyadic quality of life and dyadic relationships in lupus. Lupus. 2015 Aug;24(9):918-26. doi: 10.1177/0961203314567749. Epub 2015 Feb 5. PMID 25661509
- [Background] Israelsson J, Persson C, Bremer A, Stromberg A, Arestedt K. Dyadic effects of type D personality and perceived control on health-related quality of life in cardiac arrest survivors and their spouses using the actor-partner interdependence model. Eur J Cardiovasc Nurs. 2020 Apr;19(4):351-358. doi: 10.1177/1474515119890466. Epub 2019 Nov 22. PMID 31752502
- [Background] Boehmer U, Stokes JE, Bazzi AR, Clark MA. Dyadic quality of life among heterosexual and sexual minority breast cancer survivors and their caregivers. Support Care Cancer. 2020 Jun;28(6):2769-2778. doi: 10.1007/s00520-019-05148-7. Epub 2019 Nov 14. PMID 31724075
- [Background] Barata NE. Dyadic Relationship and Quality of Life Patients with Chronic Kidney Disease. J Bras Nefrol. 2015 Jul-Sep;37(3):315-22. doi: 10.5935/0101-2800.20150051. English, Portuguese. PMID 26398641
- [Background] Lau BH, Wong DFK, Fung YL, Zhou J, Chan CLW, Chow AYM. Facing death alone or together? Investigating the interdependence of death anxiety, dysfunctional attitudes, and quality of life in patient-caregiver dyads confronting lung cancer. Psychooncology. 2018 Aug;27(8):2045-2051. doi: 10.1002/pon.4773. Epub 2018 Jun 14. PMID 29785836
- [Background] Al-Rawashdeh S, Alshraifeen A, Rababa M, Ashour A. Hope predicted quality of life in dyads of community-dwelling patients receiving hemodialysis and their family caregivers. Qual Life Res. 2020 Jan;29(1):81-89. doi: 10.1007/s11136-019-02378-4. Epub 2019 Dec 2. PMID 31792798
- [Background] Sterba KR, Zapka J, Cranos C, Laursen A, Day TA. Quality of Life in Head and Neck Cancer Patient-Caregiver Dyads: A Systematic Review. Cancer Nurs. 2016 May-Jun;39(3):238-50. doi: 10.1097/NCC.0000000000000281. PMID 26121180
- [Background] Santos M, Sousa C, Pereira M, Pereira MG. Quality of life in patients with multiple sclerosis: A study with patients and caregivers. Disabil Health J. 2019 Oct;12(4):628-634. doi: 10.1016/j.dhjo.2019.03.007. Epub 2019 Mar 28. PMID 31005483
- [Background] Zeren F, Gursoy E, Colak E. The Quality of Life and Dyadic Adjustment of Couples Receiving Infertility Treatment. Afr J Reprod Health. 2019 Mar;23(1):117-127. doi: 10.29063/ajrh2019/v23i1.12. PMID 31034178
- [Background] Durante A, Paturzo M, Mottola A, Alvaro R, Vaughan Dickson V, Vellone E. Caregiver Contribution to Self-care in Patients With Heart Failure: A Qualitative Descriptive Study. J Cardiovasc Nurs. 2019 Mar/Apr;34(2):E28-E35. doi: 10.1097/JCN.0000000000000560. PMID 30589655
- [Background] Pucciarelli G, Ausili D, Rebora P, Arisido MW, Simeone S, Alvaro R, Vellone E. Formal and informal care after stroke: A longitudinal analysis of survivors' post rehabilitation hospital discharge. J Adv Nurs. 2019 Nov;75(11):2495-2505. doi: 10.1111/jan.13998. Epub 2019 Apr 22. PMID 30883880
- [Background] Pucciarelli G, Lee CS, Lyons KS, Simeone S, Alvaro R, Vellone E. Quality of Life Trajectories Among Stroke Survivors and the Related Changes in Caregiver Outcomes: A Growth Mixture Study. Arch Phys Med Rehabil. 2019 Mar;100(3):433-440.e1. doi: 10.1016/j.apmr.2018.07.428. Epub 2018 Aug 18. PMID 30130516
- [Background] Pucciarelli G, Ausili D, Galbussera AA, Rebora P, Savini S, Simeone S, Alvaro R, Vellone E. Quality of life, anxiety, depression and burden among stroke caregivers: A longitudinal, observational multicentre study. J Adv Nurs. 2018 Apr 27. doi: 10.1111/jan.13695. Online ahead of print. PMID 29700840
- [Background] Pucciarelli G, Vellone E, Savini S, Simeone S, Ausili D, Alvaro R, Lee CS, Lyons KS. Roles of Changing Physical Function and Caregiver Burden on Quality of Life in Stroke: A Longitudinal Dyadic Analysis. Stroke. 2017 Mar;48(3):733-739. doi: 10.1161/STROKEAHA.116.014989. Epub 2017 Feb 14. PMID 28196939
- [Background] De Maria M, Vellone E, Ausili D, Alvaro R, Di Mauro S, Piredda M, De Marinis M, Matarese M. Self-care of patient and caregiver DyAds in multiple chronic conditions: A LongITudinal studY (SODALITY) protocol. J Adv Nurs. 2019 Feb;75(2):461-471. doi: 10.1111/jan.13834. Epub 2018 Sep 19. PMID 30168154
- [Background] Zhu W, Jiang Y. A Meta-analytic Study of Predictors for Informal Caregiver Burden in Patients With Stroke. J Stroke Cerebrovasc Dis. 2018 Dec;27(12):3636-3646. doi: 10.1016/j.jstrokecerebrovasdis.2018.08.037. Epub 2018 Sep 27. PMID 30268368
- [Background] De Maria M, Matarese M, Stromberg A, Ausili D, Vellone E, Jaarsma T, Osokpo OH, Daus MM, Riegel B, Barbaranelli C. Cross-cultural assessment of the Self-Care of Chronic Illness Inventory: A psychometric evaluation. Int J Nurs Stud. 2021 Apr;116:103422. doi: 10.1016/j.ijnurstu.2019.103422. Epub 2019 Sep 26. PMID 31791631
- [Background] Philp I, Brainin M, Walker MF, Ward AB, Gillard P, Shields AL, Norrving B; Global Stroke Community Advisory Panel. Development of a poststroke checklist to standardize follow-up care for stroke survivors. J Stroke Cerebrovasc Dis. 2013 Oct;22(7):e173-80. doi: 10.1016/j.jstrokecerebrovasdis.2012.10.016. Epub 2012 Dec 21. PMID 23265778
- [Background] Turner-Stokes L. Goal attainment scaling (GAS) in rehabilitation: a practical guide. Clin Rehabil. 2009 Apr;23(4):362-70. doi: 10.1177/0269215508101742. Epub 2009 Jan 29. PMID 19179355
- [Background] Pucciarelli G, Buck HG, Barbaranelli C, Savini S, Simeone S, Juarez-Vela R, Alvaro R, Vellone E. Psychometric Characteristics of the Mutuality Scale in Stroke Patients and Caregivers. Gerontologist. 2016 Oct;56(5):e89-98. doi: 10.1093/geront/gnw083. Epub 2016 Apr 25. PMID 27114475
- [Background] Ewing G, Brundle C, Payne S, Grande G; National Association for Hospice at Home. The Carer Support Needs Assessment Tool (CSNAT) for use in palliative and end-of-life care at home: a validation study. J Pain Symptom Manage. 2013 Sep;46(3):395-405. doi: 10.1016/j.jpainsymman.2012.09.008. Epub 2012 Dec 12. PMID 23245452
- [Background] Han B, Haley WE. Family caregiving for patients with stroke. Review and analysis. Stroke. 1999 Jul;30(7):1478-85. doi: 10.1161/01.str.30.7.1478. PMID 10390326
- [Background] Shyu YI, Chen MC, Chen ST, Wang HP, Shao JH. A family caregiver-oriented discharge planning program for older stroke patients and their family caregivers. J Clin Nurs. 2008 Sep;17(18):2497-508. doi: 10.1111/j.1365-2702.2008.02450.x. PMID 18705725
- [Background] Bull MJ, Hansen HE, Gross CR. A professional-patient partnership model of discharge planning with elders hospitalized with heart failure. Appl Nurs Res. 2000 Feb;13(1):19-28. doi: 10.1016/s0897-1897(00)80015-4. PMID 10701280
- [Background] Shannon RL, Forster A, Hawkins RJ. A qualitative exploration of self-reported unmet need one year after stroke. Disabil Rehabil. 2016 Oct;38(20):2000-7. doi: 10.3109/09638288.2015.1107784. Epub 2016 Jan 5. PMID 26733052
- [Background] Low JT, Kersten P, Ashburn A, George S, McLellan DL. A study to evaluate the met and unmet needs of members belonging to Young Stroke groups affiliated with the Stroke Association. Disabil Rehabil. 2003 Sep 16;25(18):1052-6. doi: 10.1080/0963828031000069753. PMID 12944160
- [Background] Hartke RJ, Brashler R. Assessment of the needs of the young stroke survivor. Top Stroke Rehabil. 1994 Mar;1(1):15-24. doi: 10.1080/10749357.1994.11754003. PMID 27680551
- [Background] Saito M, Tadaka E, Arimoto A. Development of a family caregiver needs-assessment scale for end-of-life care for senility at home (FADE). PLoS One. 2019 Sep 11;14(9):e0222235. doi: 10.1371/journal.pone.0222235. eCollection 2019. PMID 31509587
- [Background] Bull MJ, Hansen HE, Gross CR. Differences in family caregiver outcomes by their level of involvement in discharge planning. Appl Nurs Res. 2000 May;13(2):76-82. doi: 10.1016/s0897-1897(00)80004-x. PMID 10842903
- [Background] Almborg AH, Ulander K, Thulin A, Berg S. Discharge planning of stroke patients: the relatives' perceptions of participation. J Clin Nurs. 2009 Mar;18(6):857-65. doi: 10.1111/j.1365-2702.2008.02600.x. PMID 19239664
- [Background] Finch E, Foster M, Fleming J, Cruwys T, Williams I, Shah D, Jaques K, Aitken P, Worrall L. Exploring changing needs following minor stroke. Health Soc Care Community. 2020 Mar;28(2):347-356. doi: 10.1111/hsc.12866. Epub 2019 Sep 30. PMID 31568627
- [Background] Rothwell K, Boaden R, Bamford D, Tyrrell PJ. Feasibility of assessing the needs of stroke patients after six months using the GM-SAT. Clin Rehabil. 2013 Mar;27(3):264-71. doi: 10.1177/0269215512457403. Epub 2012 Sep 5. PMID 22952306
- [Background] Magaard G, Wester P, Levi R, Lindvall P, Gustafsson E, Nazemroaya Sedeh A, Lonnqvist M, Berggren S, Nyman K, Hu X. Identifying Unmet Rehabilitation Needs in Patients After Stroke With a Graphic Rehab-CompassTM. J Stroke Cerebrovasc Dis. 2018 Nov;27(11):3224-3235. doi: 10.1016/j.jstrokecerebrovasdis.2018.07.013. Epub 2018 Aug 8. PMID 30097401
- [Background] Ing MM, Linton KF, Vento MA, Nakagawa K. Investigation of Stroke Needs (INVISION) Study: Stroke Awareness and Education. Hawaii J Med Public Health. 2015 Apr;74(4):141-5. PMID 25954601
- [Background] Chen T, Zhang B, Deng Y, Fan JC, Zhang L, Song F. Long-term unmet needs after stroke: systematic review of evidence from survey studies. BMJ Open. 2019 May 19;9(5):e028137. doi: 10.1136/bmjopen-2018-028137. PMID 31110106
- [Background] Olaiya MT, Cadilhac DA, Kim J, Nelson MR, Srikanth VK, Andrew NE, Bladin CF, Gerraty RP, Fitzgerald SM, Phan T, Frayne J, Thrift AG; STANDFIRM (Shared Team Approach Between Nurses and Doctors for Improved Risk Factor Management) Investigators. Long-term unmet needs and associated factors in stroke or TIA survivors: An observational study. Neurology. 2017 Jul 4;89(1):68-75. doi: 10.1212/WNL.0000000000004063. Epub 2017 May 31. PMID 28566545
- [Background] Wray F, Clarke D. Longer-term needs of stroke survivors with communication difficulties living in the community: a systematic review and thematic synthesis of qualitative studies. BMJ Open. 2017 Oct 6;7(10):e017944. doi: 10.1136/bmjopen-2017-017944. PMID 28988185
- [Background] Moreland JD, Depaul VG, Dehueck AL, Pagliuso SA, Yip DW, Pollock BJ, Wilkins S. Needs assessment of individuals with stroke after discharge from hospital stratified by acute Functional Independence Measure score. Disabil Rehabil. 2009;31(26):2185-95. doi: 10.3109/09638280902951846. PMID 19903128
- [Background] Abuzinadah AR, Cooke L. Neurology Health Advocacy Curriculum: Needs Assessment, Curricular Content and Underlying Components. Can J Neurol Sci. 2017 Mar;44(2):170-176. doi: 10.1017/cjn.2016.405. Epub 2016 Nov 16. PMID 27846918
- [Background] Patchwood E, Rothwell K, Rhodes S, Batistatou E, Woodward-Nutt K, Lau YS, Grande G, Ewing G, Bowen A. Organising Support for Carers of Stroke Survivors (OSCARSS): study protocol for a cluster randomised controlled trial, including health economic analysis. Trials. 2019 Jan 7;20(1):19. doi: 10.1186/s13063-018-3104-7. PMID 30616692
- [Background] Depaul VG, Moreland JD, Dehueck AL. Physiotherapy needs assessment of people with stroke following discharge from hospital, stratified by acute functional independence measure score. Physiother Can. 2013 Summer;65(3):204-14. doi: 10.3138/ptc.2012-14. PMID 24403687
- [Background] Davoody N, Koch S, Krakau I, Hagglund M. Post-discharge stroke patients' information needs as input to proposing patient-centred eHealth services. BMC Med Inform Decis Mak. 2016 Jun 7;16:66. doi: 10.1186/s12911-016-0307-2. PMID 27267889
- [Background] McCurley JL, Funes CJ, Zale EL, Lin A, Jacobo M, Jacobs JM, Salgueiro D, Tehan T, Rosand J, Vranceanu AM. Preventing Chronic Emotional Distress in Stroke Survivors and Their Informal Caregivers. Neurocrit Care. 2019 Jun;30(3):581-589. doi: 10.1007/s12028-018-0641-6. PMID 30421266
- [Background] Lynch EA, Luker JA, Cadilhac DA, Hillier SL. Rehabilitation assessments for patients with stroke in Australian hospitals do not always reflect the patients' rehabilitation requirements. Arch Phys Med Rehabil. 2015 May;96(5):782-9. doi: 10.1016/j.apmr.2014.12.009. Epub 2014 Dec 30. PMID 25555925
- [Background] Lehnerer S, Hotter B, Padberg I, Knispel P, Remstedt D, Liebenau A, Grittner U, Wellwood I, Meisel A; BSA Long Term Care Study Group. Social work support and unmet social needs in life after stroke: a cross-sectional exploratory study. BMC Neurol. 2019 Sep 6;19(1):220. doi: 10.1186/s12883-019-1451-y. PMID 31492151
- [Background] Hall JF, Crocker TF, Clarke DJ, Forster A. Supporting carers of stroke survivors to reduce carer burden: development of the Preparing is Caring intervention using Intervention Mapping. BMC Public Health. 2019 Oct 29;19(1):1408. doi: 10.1186/s12889-019-7615-2. PMID 31664985
- [Background] Groeneveld IF, Arwert HJ, Goossens PH, Vliet Vlieland TPM. The Longer-term Unmet Needs after Stroke Questionnaire: Cross-Cultural Adaptation, Reliability, and Concurrent Validity in a Dutch Population. J Stroke Cerebrovasc Dis. 2018 Jan;27(1):267-275. doi: 10.1016/j.jstrokecerebrovasdis.2017.08.043. Epub 2017 Sep 28. PMID 28967592
- [Background] Shyu YI. The needs of family caregivers of frail elders during the transition from hospital to home: a Taiwanese sample. J Adv Nurs. 2000 Sep;32(3):619-25. doi: 10.1046/j.1365-2648.2000.01519.x. PMID 11012804
- [Background] Dulhanty LH, Hulme S, Vail A, Patel HC, Tyson SF. The self-reported needs of patients following subarachnoid hemorrhage (SAH). Disabil Rehabil. 2020 Dec;42(24):3450-3456. doi: 10.1080/09638288.2019.1595748. Epub 2019 Apr 18. PMID 30999783
- [Background] King RB, Hartke RJ, Lee J, Raad J. The stroke caregiver unmet resource needs scale: development and psychometric testing. J Neurosci Nurs. 2013 Dec;45(6):320-8. doi: 10.1097/JNN.0b013e3182a3ce40. PMID 24217142
- [Background] Kersten P, Low JT, Ashburn A, George SL, McLellan DL. The unmet needs of young people who have had a stroke: results of a national UK survey. Disabil Rehabil. 2002 Nov 10;24(16):860-6. doi: 10.1080/09638280210142167. PMID 12450462
- [Background] Cameron JI, Gignac MA. "Timing It Right": a conceptual framework for addressing the support needs of family caregivers to stroke survivors from the hospital to the home. Patient Educ Couns. 2008 Mar;70(3):305-14. doi: 10.1016/j.pec.2007.10.020. Epub 2007 Dec 21. PMID 18155388
- [Background] Lin B, Ding C, Mei Y, Wang P, Ma F, Zhang ZX. Unmet care needs of community-dwelling stroke survivors: a protocol for systematic review and theme analysis of quantitative and qualitative studies. BMJ Open. 2019 Jun 21;9(6):e029160. doi: 10.1136/bmjopen-2019-029160. PMID 31230030
- [Background] Turner GM, Mullis R, Lim L, Kreit L, Mant J. Using a checklist to facilitate management of long-term care needs after stroke: insights from focus groups and a feasibility study. BMC Fam Pract. 2019 Jan 4;20(1):2. doi: 10.1186/s12875-018-0894-3. PMID 30609920
- [Background] LoTS care LUNS study team. Validation of the longer-term unmet needs after stroke (LUNS) monitoring tool: a multicentre study. Clin Rehabil. 2013 Nov;27(11):1020-8. doi: 10.1177/0269215513487082. Epub 2013 Jun 20. PMID 23787941
- [Background] Yang WFZ, Liu J, Chan YH, Griva K, Kuparasundram S, Mahendran R. Validation of the Needs Assessment of Family Caregivers-Cancer scale in an Asian population. BMC Psychol. 2020 Aug 12;8(1):84. doi: 10.1186/s40359-020-00445-x. PMID 32787927
- [Background] Moore CG, Carter RE, Nietert PJ, Stewart PW. Recommendations for planning pilot studies in clinical and translational research. Clin Transl Sci. 2011 Oct;4(5):332-7. doi: 10.1111/j.1752-8062.2011.00347.x. PMID 22029804
- [Background] Chen HL, Liu K, You QS. Effects of couple based coping intervention on self-efficacy and quality of life in patients with resected lung cancer. Patient Educ Couns. 2017 Dec;100(12):2297-2302. doi: 10.1016/j.pec.2017.07.002. Epub 2017 Jul 8. PMID 28693921
- [Background] Bandura A. Social cognitive theory: an agentic perspective. Annu Rev Psychol. 2001;52:1-26. doi: 10.1146/annurev.psych.52.1.1. PMID 11148297
- [Background] Lyons KS, Lee CS. The Theory of Dyadic Illness Management. J Fam Nurs. 2018 Feb;24(1):8-28. doi: 10.1177/1074840717745669. Epub 2018 Jan 20. PMID 29353528
- [Background] Markle-Reid M, Valaitis R, Bartholomew A, Fisher K, Fleck R, Ploeg J, Salerno J. An integrated hospital-to-home transitional care intervention for older adults with stroke and multimorbidity: A feasibility study. J Comorb. 2020 Apr 22;10:2235042X19900451. doi: 10.1177/2235042X19900451. eCollection 2020 Jan-Dec. PMID 32363165
- [Background] Lutz BJ, Young ME, Creasy KR, Martz C, Eisenbrandt L, Brunny JN, Cook C. Improving Stroke Caregiver Readiness for Transition From Inpatient Rehabilitation to Home. Gerontologist. 2017 Oct 1;57(5):880-889. doi: 10.1093/geront/gnw135. PMID 27816914
- [Background] Reeves MJ, Hughes AK, Woodward AT, Freddolino PP, Coursaris CK, Swierenga SJ, Schwamm LH, Fritz MC. Improving transitions in acute stroke patients discharged to home: the Michigan stroke transitions trial (MISTT) protocol. BMC Neurol. 2017 Jun 17;17(1):115. doi: 10.1186/s12883-017-0895-1. PMID 28623892
- [Background] Coleman EA, Smith JD, Frank JC, Min SJ, Parry C, Kramer AM. Preparing patients and caregivers to participate in care delivered across settings: the Care Transitions Intervention. J Am Geriatr Soc. 2004 Nov;52(11):1817-25. doi: 10.1111/j.1532-5415.2004.52504.x. PMID 15507057
- [Background] Connolly T, Mahoney E. Stroke survivors' experiences transitioning from hospital to home. J Clin Nurs. 2018 Nov;27(21-22):3979-3987. doi: 10.1111/jocn.14563. Epub 2018 Jul 30. PMID 29893039
- [Background] Hirschman KB, Shaid E, McCauley K, Pauly MV, Naylor MD. Continuity of Care: The Transitional Care Model. Online J Issues Nurs. 2015 Sep 30;20(3):1. PMID 26882510
- [Background] Andrew NE, Busingye D, Lannin NA, Kilkenny MF, Cadilhac DA. The Quality of Discharge Care Planning in Acute Stroke Care: Influencing Factors and Association with Postdischarge Outcomes. J Stroke Cerebrovasc Dis. 2018 Mar;27(3):583-590. doi: 10.1016/j.jstrokecerebrovasdis.2017.09.043. Epub 2017 Oct 31. PMID 29097058
- [Background] Wang Y, Yang F, Shi H, Yang C, Hu H. What Type of Transitional Care Effectively Reduced Mortality and Improved ADL of Stroke Patients? A Meta-Analysis. Int J Environ Res Public Health. 2017 May 10;14(5):510. doi: 10.3390/ijerph14050510. PMID 28489044
- [Background] Sebern MD, Whitlatch CJ. Dyadic relationship scale: a measure of the impact of the provision and receipt of family care. Gerontologist. 2007 Dec;47(6):741-51. doi: 10.1093/geront/47.6.741. PMID 18192628
- [Background] Orsulic-Jeras S, Whitlatch CJ, Powers SM, Johnson J. A dyadic perspective on assessment in Alzheimer's dementia: Supporting both care partners across the disease continuum. Alzheimers Dement (N Y). 2020 Aug 28;6(1):e12037. doi: 10.1002/trc2.12037. eCollection 2020. PMID 32885021